CLINICAL TRIAL: NCT06446349
Title: Impact of Identification and Brief Motivational Intervention in Dispensing Pharmacies (BMI) on the Deprescription of Benzodiazepines and Related Substances in Adult Chronic Drug Users
Brief Title: Brief Motivational Intervention (BMI) on the Deprescription of Benzodiazepines and Related Substances in Adult Chronic Drug Users
Acronym: BENZ_HALTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 38RC23.0198; 2023-A01747-38 (Other: ID RCB)
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Benzodiazepine Withdrawal
Keywords: substance use disorder; community pharmacy
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Brief motivational intervention in community pharmacy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief motivational intervention (Experimental): identification followed by a brief motivational intervention in pharmacies (BMI) based on the mobilisation of patients' psychosocial skills and the integration of tools to help reduce consumption of BZD/Z prescribed over the long term (≥ 6 months).
  Interventions: Other: Brief motivational intervention
- Control (No Intervention): Standard of care in case of benzodiazepine prescription

INTERVENTIONS:
Other: Brief motivational intervention — identification followed by a brief motivational intervention in pharmacies (BMI) based on the mobilisation of patients' psychosocial skills and the integration of tools to help reduce consumption of BZD/Z prescribed over the long term (≥ 6 months).
  Arms: Brief motivational intervention

SUMMARY:
We hypothesise that a short-term intervention by dispensing pharmacists is feasible and relatively easy to implement, and that it could have an impact on the deprescribing of BZD/Z in adult patients.

Two primary objectives will be evaluated in a sequential hierarchical manner, with two primary endpoints analysed one after the other, without alpha risk adjustment, but the second can only be analysed if the null hypothesis is rejected for the first:

1. Evaluate the impact of brief motivational intervention (BMI) on reducing the daily dose of BZD/Z prescribed at 6 months (superiority hypothesis) compared with the usual practice of dispensing BZD/Z in pharmacies.
2. Evaluate the impact of BMI on clinical worsening at 6 months (non-inferiority hypothesis) in comparison with the usual practice of dispensing BZD/Z in pharmacies.

DETAILED DESCRIPTION:
In France, the prevalence of use of benzodiazepines (BZDs) and related drugs (Z-drugs: zolpidem, zopiclone) (BZD/Z) was estimated at 13.4% in 2015, and 15% of new users had a first prescription exceeding the legal duration. The increase in prescriptions has continued to grow: in the first 4 months of 2021, an increase of 1.3 million anxiolytic treatments and 580,000 hypnotic treatments was observed, with new prescriptions for these treatments increasing by 15% for anxiolytics and 26% for hypnotics over the same year. The prevalence of long-term (>6 months) BZD prescriptions varies from country to country between 6% and 15% in the general population, and is estimated to reach 22% to 55% in people aged ≥ 65 years. In France, recommendations and good practice guidelines recommend prescriptions limited to 4 weeks for hypnotic BZD/Z and 12 weeks for anxiolytic BZD. However, a recent study focusing solely on anxiolytic BZDs, carried out in patients covered by the general social security system (excluding special schemes such as self-employed workers, farmers, etc.), showed that 12.2% of women and 9.3% of men aged over 50 were prescribed for longer than the legal duration.

All countries agree on the need to limit the length of time these drugs are prescribed because of the rapid inversion of the benefit/risk ratio in the case of prolonged and continuous prescribing (rapid loss of efficacy due to the tolerance effect associated with the occurrence of adverse effects.

A number of public health initiatives have been taken in France to reduce the initiation or continued use of long-term BZD/Z prescriptions, including information for healthcare professionals about the risks, pictograms on drug packaging, directives from the health authorities, incentives offered by the Assurance Maladie and regulatory measures to control prescribing. Alongside these measures, various types of psychosocial intervention are specifically aimed at deprescribing, defined as a clinically supervised process of stopping or reducing the dose of drugs when they cause harm or when the potential risks outweigh the benefits. These strategies have been evaluated for several years, ranging from brief interventions in the form of letters, self-support manuals and targeted consultations, to more complex psychotherapeutic interventions such as cognitive behavioural therapy (CBT) or pharmacological interventions.

Although complex interventions such as structured educational programmes or 3rd wave CBT have been shown to be effective in reducing long-term BZD/Z use, particularly in the elderly, they are often too long and complex to be implemented on a large scale, particularly in primary care, and all the more so in a context of increasing shortage of specialists. Brief interventions, which are both more realistic and functional, have been shown to be effective in reducing and stopping long-term use of BZD/Z at 6 and 12 months post-intervention. At the same time, very few studies have involved the active participation of pharmacy professionals. Yet the involvement of pharmacists would optimise prescribing, and a simple psychoeducation action carried out in pharmacies would have an economic impact. With a view to the shift to ambulatory care centred on the structuring of care pathways, increasing the skills of local pharmacists, as part of a multiprofessional coordination strategy, is a response to the requirements of the law modernising the French healthcare system, while offering a simple and pragmatic intervention model for patients whose prescriptions need to be optimised.

In this study, the investigators propose to evaluate the impact of identification combined with a brief motivational intervention in pharmacies (BMI) targeting the deprescription of BZD/Z in adult patients with long-term prescriptions (≥ 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Continuous treatment (at least once daily) with BZD/Z for at least 6 months, after verification of 6 months' supply.
* Signed informed consent
* Patient able to understand the survey and complete a questionnaire in French.
* Affiliation with the French social security system

Exclusion Criteria:

* Concomitant treatment with:

  * The following oral antipsychotics: risperidone, olanzapine, aripiprazole, quetiapine, clozapine, haloperidol, flupentixol, pimozide, chlorpromazine, sulpiride, zuclopenthixol, loxapine, cyamemazine (>100mg/D), sulpiride (>150mg/D),
  * Injectable medium- and long-acting antipsychotics
  * Thymoregulatory treatment with lithium
  * Treatments for alcohol use disorders: baclofen, nalmefene, naltrexone, acamprosate, disulfiram
  * Opiate substitution treatments: buprenorphine, methadone
  * Anti-epileptic drugs
* History of convulsions or epilepsy
* History of gabaergic withdrawal accidents: delirium tremens, confusional syndrome requiring specialist treatment (hospitalisation, specialist consultation), epileptic seizures, etc.
* Patients suffering from cancer
* Persons referred to in articles L1121-5 to L1121-8 of the French Public Health Code (corresponding to all protected persons: pregnant women, women in childbirth, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to a legal protection measure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of the Daily dose of BZD/Z drug | 6 months
  Change of at least 50% of the Defined Daily Dose (DDD) initially prescribed (reduction), 6 months after the BPMI (during the last 4 weeks prior to the assessment)
Worsening of the clinical symptoms of anxiety and/or sleep disorders | 6 months
  Clinical worsening is defined as:
  * An increase in anxiety ≥ 3 points of the HAD-A sub-score (the minimum clinically significant difference being estimated at 3.2 +/- 4.
  * and/or an increase ≥ 8 points in the ISI (the minimum difference corresponding to a moderate improvement being estimated at > 7 points.

SECONDARY OUTCOMES:
change of the prescribed daily dose of BZD/Z without clinical worsening (superiority hypothesis) compared with the usual practice of dispensing BZD/Z in pharmacies | 12 months
  1. Proportion of patients with a change (reduction) of at least 50% of the initially prescribed Defined Daily Dose (DDD), without clinical worsening, during the last 4 weeks prior to assessment.
complete cessation of BZD/Z prescriptions without clinical worsening (superiority hypothesis) compared with the usual practice of dispensing BZD/Z in pharmacies | 6 months and 12 months
  Proportion of patients whose BZD/Z prescription was stopped, without clinical worsening. Discontinuation is defined as no prescriptions or dispensing identified in the last 4 weeks prior to assessment.
declared consumption compared with the usual practice of dispensing BZD/Z in pharmacies | 6 months and 12 months
  declared average daily dose consumed and the number of days without consumption during the 7 days preceding the patient's visit
anxiety symptoms | 12 months
  Worsening of anxiety at 12 months is considered to be an increase in anxiety ≥ 3 points on the Hospital anxiety and depression scale (HAD-A sub-score). HAD-A is from 0 (no anxiety) to 21(max of anxiety)
depressive symptoms | 6 and 12 months
  A worsening of depression is considered to be an increase in depression ≥ 4 points on the Hospital anxiety and depression scale (HAD-D sub-score). HAD-D is from 0 (no depression) to 21 (max of depression)
Worsening of severity of insomnia | 12 months
  A worsening of insomnia is considered to be an increase in insomnia ≥ 8 points on the Insomnia Severity Index (ISI). the score varies from 0 (no insomnia) to 21 (max of insomnia)
transfers to other addictive products or behaviours | 6 and 12 months
  Evaluation of transfers to addictive products and/or behaviours on the "drugs" version of the Addictive Behaviour Intensity Questionnaire (QMICA). The score varies from 0 (no addictive behaviour) to 210 (max of addictive behaviour)
misuse of BZD/Z | 6 and 12 months
  Assessment of misuse of BZD/Z. In the absence of a questionnaire specifically evaluating the misuse of benzodiazepine drugs, the evaluation is carried out in the form of open questions.
Adverse events description | 3, 6, 9 and 12 months
  Description of all adverse events reported by patients during study follow-up. Specific monitoring of known severe adverse events related to the reduction in BZD/Z consumption, as well as falls, is carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Lucie PENNEL, MD,PhD, Principal Investigator — University Hospital, Grenoble
Locations (20):
- France (20):
  - Pharmacie Riffard Annonay, Annonay
  - Pharmacie du Village, Auriol
  - Pharmacie des Champs Dolent, Beauvais
  - Pharmacie Troisgros, Cap-d'Ail
  - Pharmacie des Fontanilles, Castelnaudary
  - Pharmacie Dolus d'Oléron, Dolus-d'Oléron
  - Pharmacie de Dommartin, Dommartin
  - Pharmacie du Mont Guillaume, Embrun
  - Ma Pharmacie Evenos, Évenos
  - Pharmacie du Pog, Lavelanet
  - Pharmacie de Lentilly, Lentilly
  - Pharmacie Thomas, Ludres
  - Pharmacie Saint Pierre Marignane, Marignane
  - Pharmacie Milan Saint-Giniez, Marseille
  - Pharmacie de la Sèvre, Moncoutant
  - Pharmacie de St georges, Saint-Georges-de-Reineins
  - Pharmacie du Théâtre, Saint-Omer
  - Pharmacie du Château, Saint-Porchaire
  - Pharmacie Labarrière, Savigné-l'Évêque
  - Pharmacie de l'Ermitage, Villemoisson-sur-Orge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Victorri-Vigneau C, Laforgue EJ, Grall-Bronnec M, Guillou-Landreat M, Rousselet M, Guerlais M; FAN-Network; Feuillet F, Jolliet P. Are Seniors Dependent on Benzodiazepines? A National Clinical Survey of Substance Use Disorder. Clin Pharmacol Ther. 2021 Feb;109(2):528-535. doi: 10.1002/cpt.2025. Epub 2020 Sep 23. PMID 32860424
- [Background] Chapoutot M, Peter-Derex L, Bastuji H, Leslie W, Schoendorff B, Heinzer R, Siclari F, Nicolas A, Lemoine P, Higgins S, Bourgeois A, Vallet GT, Anders R, Ounnoughene M, Spencer J, Meloni F, Putois B. Cognitive Behavioral Therapy and Acceptance and Commitment Therapy for the Discontinuation of Long-Term Benzodiazepine Use in Insomnia and Anxiety Disorders. Int J Environ Res Public Health. 2021 Sep 28;18(19):10222. doi: 10.3390/ijerph181910222. PMID 34639523
- [Background] Cheng JS, Huang WF, Lin KM, Shih YT. Characteristics associated with benzodiazepine usage in elderly outpatients in Taiwan. Int J Geriatr Psychiatry. 2008 Jun;23(6):618-24. doi: 10.1002/gps.1950. PMID 18058834
- [Background] Kurko TA, Saastamoinen LK, Tahkapaa S, Tuulio-Henriksson A, Taiminen T, Tiihonen J, Airaksinen MS, Hietala J. Long-term use of benzodiazepines: Definitions, prevalence and usage patterns - a systematic review of register-based studies. Eur Psychiatry. 2015 Nov;30(8):1037-47. doi: 10.1016/j.eurpsy.2015.09.003. Epub 2015 Nov 4. PMID 26545257
- [Background] Preville M, Bosse C, Vasiliadis HM, Voyer P, Laurier C, Berbiche D, Perodeau G, Grenier S, Beland SG, Dionne PA, Gentil L, Moride Y. Correlates of potentially inappropriate prescriptions of benzodiazepines among older adults: results from the ESA study. Can J Aging. 2012 Sep;31(3):313-22. doi: 10.1017/S0714980812000232. Epub 2012 Jul 17. PMID 22800936
- [Background] Airagnes G, Lemogne C, Olekhnovitch R, Roquelaure Y, Hoertel N, Goldberg M, Limosin F, Zins M. Work-Related Stressors and Increased Risk of Benzodiazepine Long-Term Use: Findings From the CONSTANCES Population-Based Cohort. Am J Public Health. 2019 Jan;109(1):119-125. doi: 10.2105/AJPH.2018.304734. Epub 2018 Nov 29. PMID 30495993
- [Background] Vinkers CH, Olivier B. Mechanisms Underlying Tolerance after Long-Term Benzodiazepine Use: A Future for Subtype-Selective GABA(A) Receptor Modulators? Adv Pharmacol Sci. 2012;2012:416864. doi: 10.1155/2012/416864. Epub 2012 Mar 29. PMID 22536226
- [Background] Morin CM, Colecchi C, Stone J, Sood R, Brink D. Behavioral and pharmacological therapies for late-life insomnia: a randomized controlled trial. JAMA. 1999 Mar 17;281(11):991-9. doi: 10.1001/jama.281.11.991. PMID 10086433
- [Background] Holbrook AM, Crowther R, Lotter A, Cheng C, King D. The diagnosis and management of insomnia in clinical practice: a practical evidence-based approach. CMAJ. 2000 Jan 25;162(2):216-20. PMID 10674058
- [Background] Linsky A, Gellad WF, Linder JA, Friedberg MW. Advancing the Science of Deprescribing: A Novel Comprehensive Conceptual Framework. J Am Geriatr Soc. 2019 Oct;67(10):2018-2022. doi: 10.1111/jgs.16136. Epub 2019 Aug 20. PMID 31430394
- [Background] Darker CD, Sweeney BP, Barry JM, Farrell MF, Donnelly-Swift E. Psychosocial interventions for benzodiazepine harmful use, abuse or dependence. Cochrane Database Syst Rev. 2015;2015(5):CD009652. doi: 10.1002/14651858.CD009652.pub2. PMID 26106751
- [Background] Lynch T, Ryan C, Hughes CM, Presseau J, van Allen ZM, Bradley CP, Cadogan CA. Brief interventions targeting long-term benzodiazepine and Z-drug use in primary care: a systematic review and meta-analysis. Addiction. 2020 Sep;115(9):1618-1639. doi: 10.1111/add.14981. Epub 2020 Feb 11. PMID 31985127
- [Background] Riordan DO, Walsh KA, Galvin R, Sinnott C, Kearney PM, Byrne S. The effect of pharmacist-led interventions in optimising prescribing in older adults in primary care: A systematic review. SAGE Open Med. 2016 Jun 14;4:2050312116652568. doi: 10.1177/2050312116652568. eCollection 2016. PMID 27354917
- [Background] Buzancic I, Dragovic P, Pejakovic TI, Markulin L, Ortner-Hadziabdic M. Exploring Patients' Attitudes Toward Deprescribing and Their Perception of Pharmacist Involvement in a European Country: A Cross-Sectional Study. Patient Prefer Adherence. 2021 Sep 23;15:2197-2208. doi: 10.2147/PPA.S323846. eCollection 2021. PMID 34588769
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] Sommer J, Rieder-Nakhle A, Gache P. [Brief motivational interventions in primary care]. Rev Med Suisse. 2007 Sep 26;3(126):2162-6. French. PMID 17969733
- [Background] Gaume J, Grazioli VS, Paroz S, Fortini C, Bertholet N, Daeppen JB. Developing a brief motivational intervention for young adults admitted with alcohol intoxication in the emergency department - Results from an iterative qualitative design. PLoS One. 2021 Feb 8;16(2):e0246652. doi: 10.1371/journal.pone.0246652. eCollection 2021. PMID 33556153
- [Background] Pottie K, Thompson W, Davies S, Grenier J, Sadowski CA, Welch V, Holbrook A, Boyd C, Swenson R, Ma A, Farrell B. Deprescription des agonistes des recepteurs des benzodiazepines: Lignes directrices de pratique clinique fondees sur les donnees probantes. Can Fam Physician. 2018 May;64(5):e209-e224. French. PMID 29760269
- [Background] Cloatre E. Regulating Alternative Healing in France, And the Problem of 'Non-Medicine'. Med Law Rev. 2019 May 1;27(2):189-214. doi: 10.1093/medlaw/fwy024. PMID 29955872
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Ohayon MM, Caulet M, Priest RG, Guilleminault C. Psychotropic medication consumption patterns in the UK general population. J Clin Epidemiol. 1998 Mar;51(3):273-83. doi: 10.1016/s0895-4356(97)00238-2. PMID 9495693
- [Background] Neutel CI. The epidemiology of long-term benzodiazepine use. Int Rev Psychiatry. 2005 Jun;17(3):189-97. doi: 10.1080/09540260500071863. PMID 16194790
- [Background] Lagnaoui R, Depont F, Fourrier A, Abouelfath A, Begaud B, Verdoux H, Moore N. Patterns and correlates of benzodiazepine use in the French general population. Eur J Clin Pharmacol. 2004 Sep;60(7):523-9. doi: 10.1007/s00228-004-0808-2. PMID 15338086
- [Background] Olfson M, King M, Schoenbaum M. Benzodiazepine use in the United States. JAMA Psychiatry. 2015 Feb;72(2):136-42. doi: 10.1001/jamapsychiatry.2014.1763. PMID 25517224
- [Background] Clay E, Falissard B, Moore N, Toumi M. Contribution of prolonged-release melatonin and anti-benzodiazepine campaigns to the reduction of benzodiazepine and Z-drugs consumption in nine European countries. Eur J Clin Pharmacol. 2013 Apr;69(4):1-10. doi: 10.1007/s00228-012-1424-1. Epub 2012 Nov 1. PMID 23114457
- [Background] Schonfeld L, Hazlett RW, Hedgecock DK, Duchene DM, Burns LV, Gum AM. Screening, Brief Intervention, and Referral to Treatment for Older Adults With Substance Misuse. Am J Public Health. 2015 Jan;105(1):205-211. doi: 10.2105/AJPH.2013.301859. PMID 24832147
- [Background] Vicens C, Bejarano F, Sempere E, Mateu C, Fiol F, Socias I, Aragones E, Palop V, Beltran JL, Pinol JL, Lera G, Folch S, Mengual M, Basora J, Esteva M, Llobera J, Roca M, Gili M, Leiva A. Comparative efficacy of two interventions to discontinue long-term benzodiazepine use: cluster randomised controlled trial in primary care. Br J Psychiatry. 2014 Jun;204(6):471-9. doi: 10.1192/bjp.bp.113.134650. Epub 2014 Feb 13. PMID 24526745
- [Background] Ng BJ, Le Couteur DG, Hilmer SN. Deprescribing Benzodiazepines in Older Patients: Impact of Interventions Targeting Physicians, Pharmacists, and Patients. Drugs Aging. 2018 Jun;35(6):493-521. doi: 10.1007/s40266-018-0544-4. PMID 29705831
- [Background] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Background] Westbury J, Jackson S, Gee P, Peterson G. An effective approach to decrease antipsychotic and benzodiazepine use in nursing homes: the RedUSe project. Int Psychogeriatr. 2010 Feb;22(1):26-36. doi: 10.1017/S1041610209991128. Epub 2009 Oct 9. PMID 19814843
- [Background] Faure G, Letoublon C, Clouye G, Guignier M, Marty F. [Value of arteriography in injuries of the kidney. The surgeon's viewpoint]. J Radiol Electrol Med Nucl. 1976 Aug-Sep;57(8-9):669-72. No abstract available. French. PMID 978637
- [Background] Navy HJ, Weffald L, Delate T, Patel RJ, Dugan JP. Clinical Pharmacist Intervention to Engage Older Adults in Reducing Use of Alprazolam. Consult Pharm. 2018 Dec 1;33(12):711-722. doi: 10.4140/TCP.n.2018.711.. PMID 30545435
- [Background] Kreek MJ, LaForge KS, Butelman E. Pharmacotherapy of addictions. Nat Rev Drug Discov. 2002 Sep;1(9):710-26. doi: 10.1038/nrd897. PMID 12209151
- [Background] Miller WR, Rollnick S. Ten things that motivational interviewing is not. Behav Cogn Psychother. 2009 Mar;37(2):129-40. doi: 10.1017/S1352465809005128. PMID 19364414
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- [Background] Atkins L, Francis J, Islam R, O'Connor D, Patey A, Ivers N, Foy R, Duncan EM, Colquhoun H, Grimshaw JM, Lawton R, Michie S. A guide to using the Theoretical Domains Framework of behaviour change to investigate implementation problems. Implement Sci. 2017 Jun 21;12(1):77. doi: 10.1186/s13012-017-0605-9. PMID 28637486
- [Background] Yang M, Morin CM, Schaefer K, Wallenstein GV. Interpreting score differences in the Insomnia Severity Index: using health-related outcomes to define the minimally important difference. Curr Med Res Opin. 2009 Oct;25(10):2487-94. doi: 10.1185/03007990903167415. PMID 19689221
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Knisely JS, Wunsch MJ, Cropsey KL, Campbell ED. Prescription Opioid Misuse Index: a brief questionnaire to assess misuse. J Subst Abuse Treat. 2008 Dec;35(4):380-6. doi: 10.1016/j.jsat.2008.02.001. Epub 2008 Jul 26. PMID 18657935
- [Background] Seppala LJ, Wermelink AMAT, de Vries M, Ploegmakers KJ, van de Glind EMM, Daams JG, van der Velde N; EUGMS task and Finish group on fall-risk-increasing drugs. Fall-Risk-Increasing Drugs: A Systematic Review and Meta-Analysis: II. Psychotropics. J Am Med Dir Assoc. 2018 Apr;19(4):371.e11-371.e17. doi: 10.1016/j.jamda.2017.12.098. PMID 29402652
- See also: Related Info — https://www.epi-phare.fr/rapports-detudes-et-publications/covid-19-usage-des-medicaments-rapport-6
- See also: Related Info — https://www.racgp.org.au/clinical-resources/clinical-guidelines/key-racgp-guidelines/view-all-racgp-guidelines/drugs-of-dependence/part-b
- See also: Related Info — https://gmmmg.nhs.uk/wp-content/uploads/2021/08/Benzodiazepine-and-Z-drug-Resource-Pack-GMMMG-FINAL-v1-0-for-GMMMG-website.pdf
- See also: Related Info — https://www.has-sante.fr/upload/docs/application/pdf/2021-02/reco403_rapport_elaboration_2014_maj2021_alcool_cannabis_tabac_cd_2021_02_05.pdf
- See also: Related Info — https://www.rfcrpv.fr/wp-content/uploads/2022/05/rapport-IATROSTAT-version-defintiive-02-mai-2022.pdf
- See also: Related Info — https://www.alcoologie-et-addictologie.fr/index.php/aa/article/view/674
- See also: Related Info — https://www.has-sante.fr/jcms/c_2038262/fr/arret-des-benzodiazepines-et-medicaments-apparentes-demarche-du-medecin-traitant-en-ambulatoire
- See also: Related Info — https://www.equator-network.org/wp-content/uploads/2014/03/TIDieR-Checklist-Word_translation-FRENCH_Dec-2017.pdf
- See also: Related Info — https://www.has-sante.fr/jcms/c_601509/fr/modalites-d-arret-des-benzodiazepines-et-medicaments-apparentes-chez-le-patient-age